CLINICAL TRIAL: NCT07133893
Title: Effects of Transcranial Photobiomodulation and Attention Bias Modification on Anxiety Symptoms and Brain Hemodynamics
Brief Title: Transcranial Photobiomodulation in Anxiety Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00007224
Record Dates: First submitted 2025-07-24; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Symptoms of Anxiety
Keywords: Photobiomodulation; Sub-clinical anxiety; Near-infrared spectroscopy (NIRS); attention bias modification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Arm 1: attention bias assessment (ABA), transcranial photobiomodulation (tPBM) (Active Comparator): Participants will receive attention bias assessment (ABA) in conjunction with active transcranial photobiomodulation (tPBM) treatment to the forehead.
  Interventions: Behavioral: Attention bias assessment and modification; Device: Transcranial photobiomodulation
- Arm 2: attention bias assessment (ABA), sham tPBM (Sham Comparator): Participants will receive attention bias assessment (ABA) in conjunction with sham (laser light off) transcranial photobiomodulation (tPBM) treatment to the forehead.
  Interventions: Behavioral: Attention bias assessment and modification
- Arm 3: attention bias assessment and modification (ABA/ABM), transcranial photobiomodulation (tPBM) (Active Comparator): Participants will receive attention bias assessment plus attention bias modification (ABA/ABM) in conjunction with active transcranial photobiomodulation (tPBM) treatment to the forehead.
  Interventions: Behavioral: Attention bias assessment and modification; Device: Transcranial photobiomodulation
- Arm 4: attention bias assessment and modification (ABA/ABM), sham tPBM (Sham Comparator): Participants will receive attention bias assessment plus attention bias modification (ABA/ABM) in conjunction with sham (laser light off) transcranial photobiomodulation (tPBM) treatment to the forehead.
  Interventions: Behavioral: Attention bias assessment and modification

INTERVENTIONS:
Behavioral: Attention bias assessment and modification — Attention bias assessment and modification involve two versions of the dot-probe task. These tasks are based on the premise that repeated attention shifts can retrain attentional biases, with the expectation that reducing attentional bias toward threats will alleviate sub-clinical anxiety symptoms.
Device: Transcranial photobiomodulation — Participants will receive near-infrared light at 1064 nanometers to the right side of the forehead for 8 minutes. The investigators have introduced this form of transcranial photobiomodulation (tPBM) as a means of human cognitive enhancement, and as an adjunct for attention bias modification for the reduction of symptoms of depression. In the present study, the investigators wish to extend these findings to the use of attention bias modification for the reduction of sub-clinical anxiety.
  Arms: Arm 1: attention bias assessment (ABA), transcranial photobiomodulation (tPBM); Arm 3: attention bias assessment and modification (ABA/ABM), transcranial photobiomodulation (tPBM)

SUMMARY:
The investigators have previously shown that safe, non-invasive methods of brain stimulation such as the administration of transcranial infrared light can result in improvements to cognition and emotion. The investigators hypothesize that transcranial photobiomodulation (tPBM) can be used in conjunction with attention bias assessment and modification to reduce anxiety symptoms in individuals with sub-clinical anxiety.

DETAILED DESCRIPTION:
The investigators will conduct two studies: one examining the efficacy of transcranial photobiomodulation as a standalone treatment to alleviate sub-clinical anxiety symptoms and another evaluating the role of transcranial photobiomodulation as an adjunct to a form of cognitive behavioral therapy in anxiety treatment. The investigators will recruit individuals with sub-clinical anxiety and use attention bias assessment (ABA) to assess levels of anxiety, and then use attention bias modification (ABM) to reduce levels of anxiety. Brain activity will be monitored using functional near-infrared spectroscopy (fNIRS).

An online prescreen questionnaire will be used to determine participant eligibility. No medical records are accessed/obtained for verifying inclusion/exclusion criteria. Informed consent is obtained during the first in-person visit. Participants fill out questionnaires to assess their medical history and anxiety/depression symptoms. The participants then participate in either ABA or ABA/ABM while wearing the fNIRS headset before and after transcranial photobiomodulation treatment or sham. Both studies will comprise three in-person visits with an online follow-up a week later. In this single-blind, sham-controlled experiment, block randomization will be performed to minimize selection bias and allocation bias.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* State-Trait Anxiety Index (STAI) questionnaire score between 40-59 (indicates moderate sub-clinical anxiety)
* Patient Health Questionnaire (PHQ-9) score between 1-9 (indicates minimal to mild sub-clinical depression)

Exclusion Criteria:

* STAI score less than 40 or greater than 59
* PHQ-9 score greater than 9
* Medication instability (i.e., medication change within 6 weeks)
* Indicated suicidal ideation
* Currently receiving tPBM treatment
* Current pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Composite cognitive score in the dot-probe task | Visit 1 (baseline), Visit 2 (three days after Visit 1), Visit 3 (1 week after Visit 2)
  The participant pays attention to a fixation cross in the center of the screen, which is followed by the presentation of two images on the left and right of the screen. One of these new images is a "threat" image, while the other is neutral. Following each trial of stimuli presentation, a probe type ("<" vs. ">") will randomly appear in the same location previously occupied by either the threatening or neutral image and remain on the screen until the participant has responded. Participants respond to the probe type by pressing the "←" or the "→" arrow key, respectively, on the keyboard, as quickly but as accurately as possible. The probe randomly replaces the neutral or the negative stimulus with equal frequency (50/50). The single primary outcome is the composite cognitive score which is calculated on the basis of performance in this task.
Change in concentration of oxygenated hemoglobin as measured by functional near-infrared spectroscopy | Visit 1 (baseline), Visit 2 (three days after Visit 1), Visit 3 (1 week after Visit 2)
  Hemodynamic activity is assessed non-invasively using near-infrared spectroscopy. In this procedure, a participant wears an apparatus on the head which contains an array of light sources and detectors. Light is applied to the surface of the skin, and a small fraction of the light passes through the underlying tissue and reflects back to the surface, where it is detected and the number of photons at specific light wavelengths are counted by a computer. This photon count can be converted to changes in concentration of metabolic indices, such as oxygenated/deoxygenated hemoglobin.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared? Individual participant data that underlie the results reported in this study, after deidentification (text, tables, figures, and appendices).
  A data dictionary, including a description of the variables and types of data, collected for each individual, will be provided. This data will include anonymized individual participant demographic information and all outcome variables (cognitive task data, spectroscopy data).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The raw data will be made available by the researchers upon reasonable request by any qualified doctoral researcher (PhD, MD). They will be granted access by contacting the corresponding author/principal investigator (F. Gonzalez-Lima, utbrainproject@gmail.com).
  It will be made available to qualified researchers whose proposed use of the data has been approved by an independent review committee (Institutional Review Board) identified for the purpose of individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in our University's shared network drive, but without investigator support other than deposited metadata.
URL: https://labs.la.utexas.edu/gonzalez-lima/idp-plan/

REFERENCES:
- [Background] Barrett DW, Beevers CG, Gonzalez-Lima F. Augmenting Internet-Based Cognitive Behavioral Therapy for Major Depressive Disorder With Transcranial Infrared Laser Stimulation. Biol Psychiatry Glob Open Sci. 2025 Jan 9;5(2):100449. doi: 10.1016/j.bpsgos.2025.100449. eCollection 2025 Mar. PMID 39990627
- [Background] Disner SG, Beevers CG, Gonzalez-Lima F. Transcranial Laser Stimulation as Neuroenhancement for Attention Bias Modification in Adults with Elevated Depression Symptoms. Brain Stimul. 2016 Sep-Oct;9(5):780-787. doi: 10.1016/j.brs.2016.05.009. Epub 2016 May 24. PMID 27267860
- [Background] Zaizar ED, Papini S, Gonzalez-Lima F, Telch MJ. Singular and combined effects of transcranial infrared laser stimulation and exposure therapy on pathological fear: a randomized clinical trial. Psychol Med. 2023 Feb;53(3):908-917. doi: 10.1017/S0033291721002270. Epub 2021 Jul 21. PMID 34284836
- See also: Gonzalez-Lima Lab Studies — https://labs.la.utexas.edu/gonzalez-lima/